CLINICAL TRIAL: NCT02011061
Title: Prospective International Study of Coronary Substraction Using 320 Row-detector CT
Brief Title: Validation of Coronary Calcium Subtraction to Improve Diagnostic Accuracy of Coronary CT Angiography
Acronym: C-Sub320
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Klaus Fuglsang Kofoed, associate professor, Rigshospitalet, Denmark
Other Study IDs: H-3-2013-108; ZIAHL006138 (NIH)
Record Dates: First submitted 2013-12-02; First posted 2013-12-13 (Estimated); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Coronary Artery Disease
Keywords: Multidetector Computed Tomography; Coronary Stenosis; Coronary Artery Disease; Angina Pectoris
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Coronary calcium hampers accurate evaluation of the coronary arteries with coronary computed tomography angiography (CCTA). A novel approach to potentially overcome this limitation is coronary calcium subtraction.

The primary hypothesis of the study is:

- Coronary calcium subtraction CCTA will improve diagnostic accuracy as compared to conventional CCTA on a per-patient basis

DETAILED DESCRIPTION:
CCTA is a very important clinical method for the clinical evaluation of patients with chest pain of potential cardiac ischemic origin. However Coronary calcification and/or previously implanted coronary stents may limit the diagnostic accuracy of CCTA. A novel approach - coronary calcium subtraction - has been developed to potentially overcome this limitation.

* Study Objective: To assess diagnostic accuracy using coronary calcium subtraction coronary CT angiography (CCTA) as compared to conventional CCTA.
* Material and Methods: A total of 200 patients with suspected or known coronary artery disease (CAD) who have been referred for invasive coronary angiography (ICA) will prior to ICA undergo additional research CCTA with the newly developed coronary calcium subtraction protocol. Based on the coronary calcium scan (CS), coronary calcium score will be calculated according to the Agatston score. Conventional contrast enhanced CCTA studies will be analyzed for image quality and the presence and extent of coronary stenosis. Using a dedicated algorithm, subtraction will be performed on all datasets to obtain CCTA subtraction images. Subtracted images will be analyzed similar to the conventional CCTA images. ICA will serve as the gold standard. Image quality will be compared between conventional and subtracted CCTA. In addition, diagnostic accuracy in the evaluation of coronary stenosis as determined on ICA will be compared. Finally, factors influencing the performance of coronary calcium subtraction will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age > 55 Years
* Scheduled for invasive coronary angiography
* Logistically possible to perform CCTA before invasive evaluation

Exclusion Criteria:

* Known Iodine-contrast allergy
* Estimated GFR below 50 ml/min
* Atrial fibrillation or other persistence cardiac arrythmia
* Contraindication to betablockers (bronchospasm, LVEF less than 40%)
* Implanted PM or ICD
* Previous mechanical heart valve surgery
* Inability to maintain breath-hold for at least 5 sec
* Patient-related condition resulting the inability of the patient to understand the informed consent form of the study

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (N=200) referred for in hospital invasive coronary evaluation
Sampling Method: Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2013-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of Coronary Subtraction Coronary CT angiography | Within 90 days of ICA and CCTA
  Sensitivity, Specificity, Negative and Positive predictive value of Coronary Subtraction CT angiography by visual assessment to identify a >50% coronary stenosis as defined by invasive coronary angiography on a patient by patient level.

SECONDARY OUTCOMES:
Coronary CT angiography reader confidence | Within 90 days of ICA and CCTA
  Coronary CT angiography reader confidence by a 3 level visual scale assessed on CT images without and with Coronary Calcium Subtraction
Coronary stenosis severity in non-diagnostic or partially diagnostic segments by conventional CCTA | Within 90 days of ICA and CCTA
  In coronary segments deemed non-diagnostic or partially diagnostic due to calcification or coronary stents by conventional CCTA concordance of stenosis severity by Coronary Subtraction CT angiography and invasive quantitative coronary angiography is assessed
Coronary revascularization | Within 30 days after CCTA
  On a patient by patient level the ability of CCTA to predict need for coronary revascularization (PCI or CABG) is assessed using CCTA without and with coronary calcium subtraction

CONTACTS AND LOCATIONS:
Overall Officials: Klaus F Kofoed, MD, DmSc, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- National Heart, Lung and Blood Institute, Bethesda, Maryland, United States
- Department of Cardiology and Radiology, Rigshospitalet, The Heart Center, Capital Region of Copenhagen, University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Background] Abdulla J, Pedersen KS, Budoff M, Kofoed KF. Influence of coronary calcification on the diagnostic accuracy of 64-slice computed tomography coronary angiography: a systematic review and meta-analysis. Int J Cardiovasc Imaging. 2012 Apr;28(4):943-53. doi: 10.1007/s10554-011-9902-6. Epub 2011 Jun 12. PMID 21667273
- [Background] Tanaka R, Yoshioka K, Muranaka K, Chiba T, Ueda T, Sasaki T, Fusazaki T, Ehara S. Improved evaluation of calcified segments on coronary CT angiography: a feasibility study of coronary calcium subtraction. Int J Cardiovasc Imaging. 2013 Dec;29 Suppl 2:75-81. doi: 10.1007/s10554-013-0316-5. Epub 2013 Oct 25. PMID 24158235
- [Background] Fuchs A, Kuhl JT, Chen MY, Helqvist S, Razeto M, Arakita K, Steveson C, Arai AE, Kofoed KF. Feasibility of coronary calcium and stent image subtraction using 320-detector row CT angiography. J Cardiovasc Comput Tomogr. 2015 Sep-Oct;9(5):393-8. doi: 10.1016/j.jcct.2015.03.016. Epub 2015 Apr 16. PMID 26091841